CLINICAL TRIAL: NCT05835050
Title: Assessment of Serum interleukin10 Level in Patients With Immune Thrombocytopenic Purpura at Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Afndia Abdelnaeem Mahmoud, Resident at Clinical pathology department at sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-11-04
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum interleukin 10 level — b. Serum levels of IL-10 were measured using a quantitative enzyme-linked immunosorbent assay (ELISA)

SUMMARY:
Autoimmune diseases are characterized by various factors that contribute to a breakdown in self-tolerance, that is, the ability of the immune system to effectively distinguish self from non-self and to refrain from attacking self. Autoimmune diseases include a broad spectrum of disorders, such as idiopathic thrombocytopenic purpura, systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, and inflammatory bowel disease. Although significant progress has been achieved in the development of approaches to the treatment of autoimmune diseases, the etiologies, and pathogenesis of autoimmune diseases remain obscure (Tao et al., 2016) Immune thrombocytopenia (ITP) is an autoimmune bleeding disorder characterized by bleeding due to isolated thrombocytopenia with platelet count less than 100 × 109/L (Neunert et al., 2019).

ITP is classified based on course of disease into acute (3- <12 months), and chronic (≥12 months) (Provan et al., 2019). ITP usually has a chronic course in adults (Moulis et al., 2017) whereas approximately 8090% of children undergo spontaneous remission within weeks to months of disease onset (Heitink et al., 2018).

The main pathogenesis of ITP is the loss of immune tolerance to platelet auto-antigens, which results in increased platelet destruction and impaired thrombopoiesis by autoantibodies and cytotoxic T lymphocytes (CTLs) (Adiua et al., 2017).

Among these abnormalities include the increased number of the T helper 1 (Th1) cells (Panitsas et al.,2004). the decreased number or defective suppressive function of regulatory T cells (Tregs) (Yu et al., 2008) , and the

ELIGIBILITY:
Inclusion Criteria:

* Patients with platelet less than 100 × 109/L diagnosed as immune thrombocytopenia according to bone marrow findings .

Exclusion Criteria:

* Other causes of thrombocytopenia as:

  * Hypersplenism.
  * Bone marrow diseases including : aplastic anemia, leukemia and myelodysplastic syndromes.
  * patients on chemotherapy and radiation therapy for cancer management

Min Age: 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
assessment of serum interleukin 10 level in patients with ITP | 16 months
  b. Serum levels of IL-10 were measured using a quantitative enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tao JH, Cheng M, Tang JP, Liu Q, Pan F, Li XP. Foxp3, Regulatory T Cell, and Autoimmune Diseases. Inflammation. 2017 Feb;40(1):328-339. doi: 10.1007/s10753-016-0470-8. PMID 27882473
- [Background] Zhan Y, Hua F, Ji L, Wang W, Zou S, Wang X, Li F, Cheng Y. Polymorphisms of the IL-23R gene are associated with primary immune thrombocytopenia but not with the clinical outcome of pulsed high-dose dexamethasone therapy. Ann Hematol. 2013 Aug;92(8):1057-62. doi: 10.1007/s00277-013-1731-3. Epub 2013 Apr 7. PMID 23564312
- [Background] Heitink-Polle KMJ, Uiterwaal CSPM, Porcelijn L, Tamminga RYJ, Smiers FJ, van Woerden NL, Wesseling J, Vidarsson G, Laarhoven AG, de Haas M, Bruin MCA; TIKI Investigators. Intravenous immunoglobulin vs observation in childhood immune thrombocytopenia: a randomized controlled trial. Blood. 2018 Aug 30;132(9):883-891. doi: 10.1182/blood-2018-02-830844. Epub 2018 Jun 26. PMID 29945954
- [Background] Audia S, Mahevas M, Samson M, Godeau B, Bonnotte B. Pathogenesis of immune thrombocytopenia. Autoimmun Rev. 2017 Jun;16(6):620-632. doi: 10.1016/j.autrev.2017.04.012. Epub 2017 Apr 17. PMID 28428120